CLINICAL TRIAL: NCT05697432
Title: Evaluation of Oral and Dental Hygiene in Individuals With Special Needs Between 6 to 12 Years of Age
Brief Title: Orodental Hygiene in Children With Special Needs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Altinbas University (Other)
Responsible Party: Principal Investigator, Mine Tirnaksiz, Principal Investigator, Altinbas University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 81
Record Dates: First submitted 2023-01-14; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Oral Hygiene
Keywords: Disabled Children; Oral Hygiene; Streptococcus mutans
MeSH Terms: interventions — Physical Examination; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education (Experimental): The children with special needs will receive a complete oral examination and then their parent/guardian will be subjected to education about oral hygiene, brushing and dietary guidance.
  Interventions: Diagnostic Test: Oral Examination; Diagnostic Test: PUFA index; Diagnostic Test: Plaque index; Diagnostic Test: Streptococcus mutans screening; Behavioral: Education

INTERVENTIONS:
Diagnostic Test: Oral Examination — A complete examination of oral and dental hygiene any health problems will be registered
Diagnostic Test: PUFA index — An assessment of the presence of oral conditions resulting from untreated caries. P=Pulpal involvement, U=ulceration, F=fistula, A=abscess index
  Other Names: Pulpal involvement, ulceration, fistula, abscess index
Diagnostic Test: Plaque index — An assessment of the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth. The index varies between 0-4.
  Other Names: Sillness Löe PI
Diagnostic Test: Streptococcus mutans screening — A strip test for specific bacteria named streptococcus mutans, which plays an important role in caries formation, from patients' collected saliva
  Other Names: Saliva-check mutans
Behavioral: Education — Education on correct toothbrushing technique, oral hygiene, dietary education on foods detrimental for dental hygiene.

SUMMARY:
This clinical trial aims to learn about the general oral hygiene status of children with special needs and test the effect of hygiene education on their oral and dental hygiene. The main questions it aims to answer are:

* What is the general oral hygiene status of children with special needs?
* Does brushing education and dietary guidance to parents improve oral and dental hygiene in children with special needs? Participants will receive a complete oral and dental examination. Following this examination parents/legal guardians will be educated about the maintenance of oral and dental hygiene and dietary guidance will be provided. Patients will be evaluated one year after the education

DETAILED DESCRIPTION:
One hundred and thirty children with special needs who are being rehabilitated at three rehabilitation centers (Maviel, Sirinler and Ugurlu Kalpler Rehabilitation Centers) in Kilis will undergo a complete oral and dental examination at which their oral bacteria (str. mutans) levels, PUFA and plaque indexes (indices that measure oral health) will be recorded. The parents/legal guardians of the children will be educated about dental hygiene toothbrushing and dietary habits leading to caries. After a year, the examination and assessments will be repeated. The change in oral hygiene indices will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children with special needs
* Aged between 6-12 years

Exclusion Criteria:

* Refusal
* Being unable to complete oral examination due to lack of cooperation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Saliva Check mutans test at 52 weeks | Baseline and 1 year after the education
  A speed test of specific bacteria named streptococcus mutans, which plays a leading role in caries formation, from patients' collected saliva. Interpreted from the strips as high, low levels of bacteria or no bacteria in saliva.
Change from baseline in the number of teeth with each element of PUFA index at 52 weeks | Baseline and 1 year after the education
  An assessment of the presence of oral conditions resulting from untreated caries. P=Pulpal involvement, U=ulceration, F=fistula, A=abscess index.
Change from baseline on the 5 point plaque index at 52 weeks | Baseline and 1 year after the education
  An assessment of the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth. Possible scores range from 0 (no plaque) to 4 (considerable plaque film formation)

CONTACTS AND LOCATIONS:
Overall Officials: Mine Tirnaksiz, Principal Investigator — Altinbas University
Locations (3):
- Turkey (Türkiye) (3):
  - Maviel Rehabilitation Center, Kilis
  - Sirinler Rehabilitation Center, Kilis
  - Ugurlu Kalpler Rehabilitation Center, Kilis

IPD SHARING:
Plan to Share IPD: No